CLINICAL TRIAL: NCT03784482
Title: Multiple Drug Hypersensitivity Syndrome in a Large Database
Brief Title: Multiple Drug Hypersensitivity Syndrome
Acronym: MDH
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0478
Record Dates: First submitted 2018-12-10; First posted 2018-12-24 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Drug Allergy
Keywords: Multiple Drug Hypersensitivity; drug hypersensitivity; antibiotics; drug provocation tests; skin tests
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Multiple drug hypersensitivity syndrome (MDH) is defined as confirmed drug hypersensitivity reactions (DHRs) to at least 2 chemically and pharmacologically unrelated drugs. Reports of MDH are scarce and poorly specified and studies which diagnose MDH on the basis of positive allergy tests are lacking.

Objective: To evaluate retrospectively the frequency and characteristics of MDH patients in a large database.

Methods: All the patients who consulted and were tested in our Allergy Unit between September 1996 and February 2018, with confirmed MDH will be included. Clinical history and allergy work-up results will be extracted from our Drug Allergy and Hypersensitivity Database (DAHD). The frequency of MDH will be calculated, MDH patients will be described, the most frequent associations of DHRs will be identified and analysed.

ELIGIBILITY:
Inclusion criteria:

* Patients who consulted at our allergy clinic (University Hospital of Montpellier, France)
* Between September 1996 and February 2018 with a clinical history suggestive of DHR
* Who completed a tailored drug allergy work-up, (including a drug allergy questionnaire, skin tests (STs) and drug provocation tests (DPTs)) and were diagnosed with MDH.

Exclusion criteria:

* the DHR was due to a single component contained in 2 different drug formulations
* in composed drugs;
* there was possible cross-reactivity between the responsible drugs; (iv) the patient had positive but non standardized nor validated (i.e. possibly irritant)
* these STs were followed by a negative DPT;
* DPTs with placebo were positive; (vii) doubtful tests were repeated and eventually considered negative;
* a single DHR was associated with one or more non-drug related contact allergies;
* DPTs elicited subjective manifestations (i.e., isolated pruritus, headache, isolated abdominal pain);
* non-specific histamine release was suspected (e.g., chronic spontaneous - desensitization, rather than a diagnostic work-up was preferred in order to meet the urgent therapeutic needs of individual patients (HIV infected patients, cardiac patients).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient consulting in our allergy unit for a suspicion of drug hypersensitivity and who underwent diagnostic drug allergy testing
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
To measure retrospectively the frequency of MDH patients in our database. | 1 day
  The frequency of MDH patients (percentage) in the allergic group of patients will be calculated as the number of MDH patients divided by the number of monoallergic patients (frequency of MDH patients in allergic population)
To measure retrospectively the frequency of MDH patients in our database | 1 day
  The frequency of MDH in common population will be calculated by will be calculated as the number of MDH patients divided by the number of patients that underwent diagnostic drug allergy testing within the same time frame (frequency of MDH patients in the whole population

SECONDARY OUTCOMES:
To describe the MDH population, identify the most frequent associations of DHR | 1 day
  In this MDH patients population we will : Count the number of female and male patient according to their sex (No unit)
To describe the MDH population, identify the most frequent associations of DHR | 1 day
  In this MDH patients population we will : Most frequent associations of DHR (No unit)
To describe the MDH population, identify the most frequent associations of DHR | 1 day
  In this MDH patients population we will : Count and classify the different form of DHR according to their severity with the Ring and Messsmer and Regiscar study group scoring. (No unit) (ex: number of patient with grade III anaphylaxis or number of patient with DRESS syndrome )

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DEMOLY, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No